CLINICAL TRIAL: NCT00664144
Title: Study of Efficacy and Safety of Rasburicase for the Treatment/Prevention of Hyperuricemia Related to Tumor Lysis Syndrome in Adult Patients With Relapsing Aggressive Non Hodgkin's Lymphoma, Previously Treated or Not With Urate Oxidase Presenting With Hyperuricemia and/or Bulky Disease
Brief Title: Rasburicase for the Treatment/Prevention of Hyperuricemia in Adult Patients With Relapsing Aggressive Non Hodgkin's Lymphoma
Acronym: GRAAL2
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: due to poor enrollment
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, Sanofi-aventis
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: EFC4983; L_8433
Record Dates: First submitted 2008-04-18; First posted 2008-04-22 (Estimated); Last update posted 2012-03-07 (Estimated); Status verified 2012-03

CONDITIONS: Hyperuricemia
MeSH Terms: conditions — Hyperuricemia | interventions — rasburicase; Urate Oxidase

INTERVENTIONS:
Drug: Rasburicase (SR29142)

SUMMARY:
The primary objective was to evaluate the efficacy of rasburicase in terms of prevention and treatment of hyperuricemia related to Tumor Lysis Syndrome (TLS) in 2 populations of adult patients, previously treated or not with urate oxidase, with relapsing aggressive non-Hodgkin's lymphoma (NHL) and at risk of TLS, presenting with hyperuricemia and/or bulky disease at diagnostic of relapse.

The secondary objectives were to :

* evaluate the efficacy of rasburicase in terms of renal protection,
* evaluate the safety of rasburicase in the two cohorts of patients,
* correlate efficacy and safety results with antibodies generation/level.

ELIGIBILITY:
Patients with histologically proven aggressive Non Hodgkin's Lymphoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2002-07; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
responder rate (based on normalization of uric acid levels)

CONTACTS AND LOCATIONS:
Overall Officials: ICD, Study Director — Sanofi
Locations (4):
- Sanofi-Aventis Administrative Office, Diegem, Belgium
- Sanofi- Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Berlin, Germany
- Sanofi-Aventis Administrative Office, Milan, Italy